CLINICAL TRIAL: NCT03308123
Title: PERFECTED WP1 P4: A Qualitative Exploration of Lay and Professional Stakeholder Views of Care Delivery in Hospitals for Patients With Hip-fracture & Memory Difficulties
Brief Title: PERFECTED: Caring for Patients With Hip-fracture & Memory Difficulties
Acronym: PERFECTED
Status: Completed | Type: Observational
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Other Study IDs: 15/EE/0007; DTC-RP-PG-0311-12004 (Other Grant/Funding Number: National Institute for Health Research)
Record Dates: First submitted 2017-08-09; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-08

CONDITIONS: Dementia; Hip Fractures
MeSH Terms: conditions — Dementia; Hip Fractures | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Health Care Professionals: Health care professionals
  Interventions: Other: Observational study, not interventional
- Carers of hip-fracture patients with moderate/severe: Carers of hip-fracture patients with moderate/severe
  Interventions: Other: Observational study, not interventional
- Discharged hip-fracture patient with memory difficulty: Discharged hip-fracture patient with memory difficulty
  Interventions: Other: Observational study, not interventional

INTERVENTIONS:
Other: Observational study, not interventional — Not an intervention study

SUMMARY:
This qualitative study is part of the 5-year long (2013-18) PERFECTED (Peri-operative Enhanced Recovery hip-fracture Care of paTiEnts with Dementia) National Institute for Health Research (NIHR) funded research programme. PERFECTED's overall aim is to develop and pilot an evidence-based intervention to improve the hospital care of patients living with dementia who have fractured their hip. The findings from this particular study will support PERFECTED's other activities by exploring stakeholder (lay and professional) views of the hospital care experiences of hip-fracture patients who are experiencing memory difficulties. Best practices and priorities, including attention to cost-consequences will be explored.

Semi-structured interviews will be conducted with 15-30 hip-fracture patients with mild memory difficulties recently discharged from acute hospitals in Norwich, Nottingham and Bradford. Equal attention will be given to those patients discharged directly home and those discharged to community hospitals for further rehabilitation. Interviews will be conducted with 15-30 recognised carers of hip-fracture patients with moderate/severe memory difficulties who have recently been discharged from acute hospitals in the same three regions. Semi-structured interviews will also be carried out with a nominated dementia lead in each region. Finally, in each region, small focus groups, face-to-face or telephone interviews will be conducted, with clinical staff of various grades and professions, hospital managers and with NHS commissioners. This study will enable a range of topics and perspectives to be explored and potential components for PERFECTED's intervention to be identified.

As part of PERFECTED's on-going commitment to Public Patient Involvement (PPI), lay researchers will be trained to assist in interviewing recognised carers of hip-fracture patients with moderate/severe memory difficulties. Interviews and focus groups will be recorded, transcribed and analysed thematically. Resulting data will address the pre-defined aims of the current study and feed into findings reported across the whole of Work Package 1 of PERFECTED.

ELIGIBILITY:
Inclusion Criteria:

* A hip-fracture patient recently discharged (within a month) from an acute hospital in one of the study locations.
* 60 years or older
* Having some memory difficulties as recognised by a relevant member of their care team - supported by an AMT score of 5-8 if required
* Has the cognitive ability to engage with a research interview as determined by a relevant member of their care team

Exclusion Criteria:

* Lacks mental capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recently discharged (within a month) hip-fracture patients with mild memory difficulties
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2016-02-22 (Actual)

PRIMARY OUTCOMES:
Semi-Structure Interview | 1 month
  Stakeholder experiences

CONTACTS AND LOCATIONS:
Overall Officials: George C Fox, Principal Investigator — University of East Anglia
Locations (1):
- University of East Anglia, Norwich, Norfolk, United Kingdom